CLINICAL TRIAL: NCT06881277
Title: Effectiveness of a Smartphone App (PRIMI) to Promote Healthy Diet and Physical Activity After Pregnancy in Migrant Women
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Linkoeping University (Other Government)
Responsible Party: Principal Investigator, Pontus Henriksson, Principal Investigator, Linkoeping University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 2022-06733-01
Record Dates: First submitted 2025-03-06; First posted 2025-03-18 (Actual); Last update posted 2025-09-16 (Actual); Status verified 2025-09

CONDITIONS: Postpartum
Keywords: mHealth; app; randomized controlled trial; postpartum; pregnancy; migration; migrant health; diet; physical activity; health literacy
MeSH Terms: conditions — Alzheimer Disease; Motor Activity

STUDY DESIGN:
Who Masked: Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intervention group (Access to the PRIMI app + standard care) (Experimental): Participants randomized to the intervention group will receive standard postpartum care plus access to the PRIMI app for 6 months. The PRIMI app is a mobile health (mHealth) intervention designed to promote healthy dietary habits, physical activity, and health literacy among migrant women after pregnancy
  Interventions: Behavioral: Mobile phone based intervention
- Control group (standard care) (No Intervention): Participants in the control group will receive standard postpartum care. After the six-month follow-up, they will be granted access to the PRIMI app (wait-list control).

INTERVENTIONS:
Behavioral: Mobile phone based intervention — The PRIMI intervention is a 6-month smartphone-based digital health program designed to promote a healthy diet and physical activity among migrant women after pregnancy.
  Arms: Intervention group (Access to the PRIMI app + standard care)

SUMMARY:
The PRIMI trial (Promoting Reproductive health In MIgrant women) is a randomized controlled trial evaluating the effectiveness of a smartphone app designed to promote a healthy diet, physical activity, and health literacy among first-generation migrant women after pregnancy. The study will recruit 200 women within six months after pregnancy and randomize them into an intervention group, receiving access to the PRIMI app for six months, or a wait-list control group. The primary outcomes are diet quality and moderate-to-vigorous physical activity, while secondary outcomes include health literacy, body mass index, self-efficacy, and self-rated health. The intervention is expected to provide accessible and culturally tailored support to improve postpartum health behaviors.

DETAILED DESCRIPTION:
1. BACKGROUND

   International migrants represent a growing population in Sweden and many European countries. Currently, approximately 25% of women of childbearing age in Sweden have migrated (hereafter referred to as "migrant women"). Evidence suggests that migrant women face a higher risk of adverse health outcomes during and after pregnancy. Thus, improving migrant health, including reproductive health, is a public health priority. The period after pregnancy presents a critical opportunity to promote healthy dietary habits, physical activity, and body weight. However, there is a lack of lifestyle interventions after pregnancy tailored specifically for migrant women. Mobile health (mHealth) interventions are potentially effective in this regard, given that mobile phones are widely accessible across different socioeconomic groups. Previous research has demonstrated the potential of mHealth interventions to improve diet and physical activity. However, no previous study has evaluated the effectiveness of an mHealth intervention on health behaviors and body weight among migrant women after pregnancy.

   The PRIMI project (Promoting Reproductive Health In MIgrant Women) aims to address this gap by assessing the effectiveness of a smartphone app to support healthy behaviors after pregnancy in migrant women. The PRIMI trial will evaluate the effectiveness of a smartphone app (PRIMI app) on: i) Diet quality (primary outcome) ii) Moderate-to-vigorous physical activity (primary outcome) iii) Health literacy (secondary outcome) iv) Body mass index (BMI) (secondary outcome) v) Self-efficacy (secondary outcome) vi) Self-rated health (secondary outcome)
2. METHODS

2.1 Study Design

The PRIMI trial is a 6-month, two-arm randomized controlled trial (RCT) with a 1:1 allocation ratio. The intervention group will receive standard postpartum care plus access to the PRIMI app for six months. The control group will receive standard postpartum care and will gain access to the PRIMI app after the six-month follow-up (wait-list control design). The study follows the SPIRIT 2013 guidelines and will be reported according to the CONSORT-EHEALTH checklist.

2.2 Eligibility and Recruitment

Participants will be recruited through maternal and child healthcare services across Sweden. If recruitment is slow, additional strategies, such as outreach through non-governmental organizations, community associations, and social media, will be considered.

2.3 Randomization and Blinding

Participants will be randomly assigned to the intervention or control group using a 1:1 allocation ratio. Allocation will be concealed.

2.4 The PRIMI app

The PRIMI app consists of a 6-month structured program with weekly themes, goal-setting features, self-monitoring tools, and an extensive library of recipes, exercise videos, and behavior change support. The intervention is based on social cognitive theory and incorporates behavior change techniques such as shaping knowledge, feedback and monitoring, and goal setting. The app provides culturally adapted dietary and physical activity guidelines based on current recommendations and includes multimedia elements (e.g., images, audio, and video) for accessibility.

ELIGIBILITY:
Inclusion Criteria:

* First-generation migrant women
* Given birth ≤ 6 months ago
* Age ≥ 18 years
* Able to receive health-related information in Arabic, Somali, English, or Swedish

Exclusion Criteria:

* Swedish-born women
* Age < 18 years
* Given birth > 6 months ago

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2025-09-15 (Estimated); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Diet quality | Baseline and 6 months post-randomization.
  Assessed using a modified version of the Swedish National Board of Health and Welfare's dietary survey. A composite dietary quality score will be created based on intakes of: i) vegetables, ii) fruits and berries, iii) sweet beverages, and iv) sweet and savory snacks.
Moderate-to-vigorous physical activity | Baseline and 6 months post-randomization.
  Assessed via self-reported time spent in moderate and vigorous physical activity per day using a modified version of the physical activity questions in the Swedish National Board of Health and Welfare's survey.

SECONDARY OUTCOMES:
Dietary intakes | Baseline and 6 months post-randomization.
  Assessed using a modified version of the Swedish National Board of Health and Welfare's dietary survey. In addition to the composite diet quality score, we will examine the effectiveness of the PRIMI app on the four key indicators individually: i) vegetables, ii) fruit and berries, iii) sweet beverages, iv) sweet and savory snacks.
Physical activity | Baseline and 6 months post-randomization.
  Assessed using a modified version of the physical activity questions in the Swedish National Board of Health and Welfare's survey. Beyond analyzing the effects on moderate-to-vigorous physical activity, we will also assess moderate and vigorous physical activity separately.
Health literacy | Baseline and 6 months post-randomization.
  Measured using the Health Literacy Survey Questionnaire-16 (HLS-Q16). Scores range from 16 to 64, with higher scores indicating higher health literacy.
eHealth literacy | Baseline and 6 months post-randomization.
  Measured using the eHealth Literacy Scale (eHEALS). Scores range from 8 to 40, with higher scores indicating higher eHealth literacy.
Body mass index (BMI) | Baseline and 6 months post-randomization.
  Calculated from self-reported weight and height (kg/m²).
Self-efficacy | Baseline and 6 months post-randomization.
  Measured using a questionnaire regarding participants' perceived self-efficacy in having a healthy diet and physical activity. Scores range from 0 (not at all) to 10 (very much), with higher scores indicating greater perceived self-efficacy regarding healthy diet and physical activity.
Self-rated health | Baseline and 6 months post-randomization.
  Assessed using the EQ-5D Visual Analogue Scale (EQ-VAS). The EQ-5D VAS ranges from 0 (worst imaginable health state) to 100 (best imaginable health state). Thus, higher scores indicate better self-rated health

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Seitero A, Shirvanifar M, Jubran Leksell M, Rydfjord M, Al-Saedi B, Salah Ahmed A, Gharakhani Bahar T, Berglind D, Henriksson H, H Ahlqvist V, Wangdahl J, Mussener U, Henriksson P. A Smartphone App (PRIMI) to Promote Healthy Diet, Physical Activity, and Health Literacy After Childbirth Among Migrant Women: Protocol for a Randomized Controlled Trial. JMIR Res Protoc. 2025 Oct 17;14:e79277. doi: 10.2196/79277. PMID 41106816